CLINICAL TRIAL: NCT03379428
Title: Phase I/II Trial of Ibrutinib Plus Trastuzumab in HER2-amplified Metastatic Breast Cancer
Brief Title: Trial of Ibrutinib Plus Trastuzumab in HER2-amplified Metastatic Breast Cancer
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: US Oncology Research (Industry)
Collaborators: AbbVie (Industry); Pharmacyclics LLC. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 14059; 14-059 (Other: US Oncology Research/McKesson Specialty Health, Inc.)
Record Dates: First submitted 2017-12-12; First posted 2017-12-20 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Breast Neoplasms; Malignant Neoplasm of Breast
Keywords: Breast Cancer; Metastatic Breast Cancer; HER2-amplified Metastatic Breast Cancer; HER2-positive Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Trastuzumab; ibrutinib

STUDY DESIGN:
Intervention Model Description: This is a Phase I/II, open-label, unblinded, nonrandomized, standard 3+3 dose-escalation study designed to evaluate the maximum tolerated dose (MTD) and dose-limiting toxicities (DLT) of ibrutinib (560 or 840 or 420 mg QD) given orally in combination with trastuzumab (8 mg/kg loading dose followed by 6 mg/kg q3w) administered intravenously (IV) in patients with HER2-amplified MBC.
  Once the recommended phase II dose of ibrutinib plus trastuzumab has been determined (no more than 1 of 6 patients with dose-limiting toxicity) in the required 6 to 18 patients over the 3 possible dose levels, additional patients will be enrolled on the phase II part of the study at the recommended phase II dose of ibrutinib plus trastuzumab, for a maximum of 51 patients total.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Trastuzumab plus Ibrutinib 560 mg (Experimental): In Phase I, starting dose of Ibrutinib will be 560 mg orally per day. 3 patients will be enrolled first. If none of these have DLTs, 3 new patients will be enrolled at the next higher Ibrutinib dose level (840 mg orally per day). If 1 of these 3 patients have a DLT, expand this arm to 6 patients. If 2 or more of these 6 patients have a DLT, enroll 3 patients in lower dose lever (420 mg).
  Interventions: Drug: Trastuzumab; Drug: Ibrutinib 560 mg
- Trastuzumab plus Ibrutinib 840 mg (Experimental): If no patients in 560 mg arm have DLTs, this arm will be opened in Phase I to see how this higher dose is tolerated.
  Interventions: Drug: Trastuzumab; Drug: Ibrutinib 840 mg
- Trastuzumab plus Ibrutinib 420 mg (Experimental): If 2 or more patients in 560 mg arm have DLTs, this arm will be opened in Phase I to see how this lower dose is tolerated.
  Interventions: Drug: Trastuzumab; Drug: Ibrutinib 420 mg
- Phase II- Trastuzumab plus Maximum Tolerated Dose (Experimental): Maximum tolerated dose from Phase I will be used here in Phase II.
  Interventions: Drug: Trastuzumab

INTERVENTIONS:
Drug: Trastuzumab — 8 mg/kg loading dose (first dose), followed by 6 mg/kg every 3 weeks, administered intravenously (IV)
  Other Names: Herceptin
Drug: Ibrutinib 560 mg — 560 mg by mouth daily
  Other Names: Imbruvica; PCI-32765
  Arms: Trastuzumab plus Ibrutinib 560 mg
Drug: Ibrutinib 840 mg — 840 mg by mouth daily
  Other Names: Imbruvica; PCI-32765
  Arms: Trastuzumab plus Ibrutinib 840 mg
Drug: Ibrutinib 420 mg — 420 mg by mouth daily
  Other Names: Imbruvica; PCI-32765
  Arms: Trastuzumab plus Ibrutinib 420 mg

SUMMARY:
This is a Phase I/II, open-label dose-escalation study designed to evaluate the maximum tolerated dose (MTD) and dose-limiting side effects of ibrutinib (560 or 840 or 420 mg daily oral dose), given in combination with trastuzumab administered through the vein, in patients with HER2-amplified Metastatic Breast Cancer that has gotten worse after prior therapy with ado-trastuzumab emtansine (T-DM1).

DETAILED DESCRIPTION:
Ado-trastuzumab emtansine (T-DM1) is approved by the FDA for patients with HER2-positive metastatic breast cancer (MBC) previously treated with a taxane and trastuzumab, and is currently listed as the preferred second-line therapy in the NCCN guidelines (NCCN 2014). While the benefit of continued HER2 inhibition has been conclusively established for disease that has progressed on a trastuzumab-containing regimen, there are currently no data regarding the efficacy of HER2- targeted therapies following progression on T-DM1.

With the population of T-DM1-treated patients steadily growing, clinical trials are needed to investigate novel therapies in this setting,to meet the medical need for effective, evidence-based therapies for these patients.

The oral small-molecule Bruton's Tyrosine Kinase (BTK) inhibitor ibrutinib has also demonstrated the ability to inhibit erythroblastosis virus oncogene B (ErbB)/HER receptor family kinases in preclinical studies at clinically relevant concentrations, with an equivalent or greater potency than other HER2-directed tyrosine kinase inhibitors (TKIs) with demonstrated activity in HER2-positive MBC, including lapatinib, neratinib, and afatinib. Of note, in preclinical HER2-positive cell model systems the growth inhibitory ability of ibrutinib was substantially greater in HER2-amplified breast cancer cells versus those that simply overexpressed the HER2 protein.

Ibrutinib is currently approved for use in patients with Chronic lymphocytic leukemia (CLL) or Mantle cell lymphoma (MCL), and has an established safety record from clinical trials in these patient populations. Thus there is a reasonable rationale to investigate ibrutinib in patients with HER2- amplified MBC, in the setting of T-DM1-pretreated disease. Previous studies have demonstrated that combined targeting of HER2 with multiple HER2-directed agents is more effective that single agent therapy and therefore this study will explore the safety and efficacy of ibrutinib in combination with trastuzumab.

This is a Phase I/II, open-label, unblinded, nonrandomized, standard 3+3 dose-escalation study designed to evaluate the maximum tolerated dose (MTD) and dose-limiting toxicities (DLT) of ibrutinib (560 or 840 or 420 mg QD) given orally in combination with trastuzumab (8 mg/kg loading dose followed by 6 mg/kg q3w) administered intravenously (IV) in patients with HER2-amplified MBC that has progressed on prior therapy with ado-trastuzumab emtansine.

Once the recommended phase II dose of ibrutinib plus trastuzumab has been determined (no more than 1 of 6 patients with dose-limiting toxicity) in the required 6 to 18 patients over the 3 possible dose levels, additional patients will be enrolled on the phase II part of the study at the recommended phase II dose of ibrutinib plus trastuzumab, for a maximum of 51 patients total.

ELIGIBILITY:
Inclusion Criteria:

* 1. Female, Age ≥ 18 years
* 2. Histologic or cytologic confirmation of HER2-amplified breast cancer according to most recent biopsy (local testing permitted)

  * a. HER2-amplified status is defined as a HER2/CEP17 ratio ≥2 or an average of ≥6 HER2 gene copies per cell by in situ hybridization (ISH) according to the 2013 American Society of Clinical Oncology (ASCO)/CAP guidelines
* 3. Measurable or evaluable metastatic disease by RECIST (v1.1).
* 4. Progression of disease on or ≤6 months of completing prior TDM1 therapy
* 5. ≤ 4 prior chemotherapy regimens for MBC (Phase I portion) or ≤ 3 prior chemotherapy regimens for MBC (Phase II portion)
* 6. Adequate hematologic function independent of transfusion and growth factor support for ≤7 days prior to screening, with the exception of pegylated G-CSF (pegfilgrastim) and darbepoetin which require discontinuation at least 14 days prior to screening, defined as:

  * Absolute neutrophil count >1500 cells/mm3 (0.75 x 10^9/L).
  * Platelet count >100,000 cells/mm3 (50 x 10^9/L).
  * Hemoglobin >9.0 g/dL.
* 7. Adequate hepatic and renal function defined as:

  * Serum aspartate transaminase (AST) and/or alanine transaminase (ALT) ≤5.0 x upper limit of normal (ULN) if liver metastases, or ≤3 x ULN in the absence of liver metastases.
  * Alkaline phosphatase <2.5 x ULN, unless bone metastases are present and in the absence of liver metastases
  * Estimated Creatinine Clearance ≥30 ml/min (Cockcroft-Gault)
  * Bilirubin ≤1.5 x ULN (unless bilirubin rise is due to Gilbert's syndrome or of non-hepatic origin, such as hemolysis)
* 8. Prothrombin time (PT)/international normalized ratio (INR) < 1.5xULN and PTT (aPTT) < 1.5x ULN
* 9. Left Ventricular Ejection Fraction (LVEF) ≥ 50% at baseline as determined by either ECHO or multiple gated acquisition scan (MUGA) and within normal limits per institutional guidelines
* 10. Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2.
* 11. Negative urine/serum pregnancy test within 72 hours before starting study medications for women of childbearing potential
* 12. Women of childbearing potential who agree to use two highly effective methods of birth control (e.g., some intrauterine devices [IUD], diaphragm with spermicide, condom with spermicide, sterilized partner, or complete abstinence) for the duration of the study and for 30 days after the last dose of study drug

  o Note: Women are considered postmenopausal and not of childbearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g. age appropriate, history of vasomotor symptoms), or if they have undergone surgical sterilization
* 13. Signed informed consent obtained prior to any screening procedures.
* 14. Signed Patient Authorization Form (HIPAA) obtained prior to any screening procedures.

Exclusion Criteria:

* 1. Uncontrolled or untreated central nervous system metastases, defined as clinical or radiologic evidence of progression of brain metastases or clinical signs of leptomeningeal disease

  1. Patients with treated brain metastases are eligible provided they do not have clinical or radiologic evidence of disease progression and have been off of dexamethasone for ≥2 weeks prior to first dose of study drugs
  2. Brain MRI at baseline required for patients with known brain metastases at study entry
* 2. Chemotherapy ≤ 21 days prior to first administration of study treatment
* 3. History of other malignancies, except:

  * Malignancy treated with curative intent and with no known active disease present for ≥3 years before the first dose of study drug and felt to be at low risk for recurrence by treating physician.
  * Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease.
  * Adequately treated carcinoma in situ without evidence of disease.
* 4. Concurrent systemic immunosuppressant therapy (e.g., cyclosporine A, tacrolimus, etc., or chronic administration days] [ > 14 days] of >5 mg/day of prednisone) ≤28 days of the first dose of study drug.
* 5. Vaccinated with live, attenuated vaccines ≤4 weeks of first dose of study drug.
* 6. Recent infection requiring systemic treatment that was completed ≤14 days before the first dose of study drug.
* 7. Unresolved toxicities from prior anti-cancer therapy, defined as having not resolved to Common Terminology Criteria for Adverse Event (CTCAE, version 4), grade 0 or 1, or to the levels dictated in the inclusion/exclusion criteria with the exception of alopecia.
* 8. Known bleeding disorders (e.g., von Willebrand's disease) or hemophilia.
* 9. History of stroke or intracranial hemorrhage ≤6 months prior to first dose of study drug.
* 10. Known history of human immunodeficiency virus (HIV) or active with hepatitis C virus (HCV) or hepatitis B virus (HBV). Patients who are positive for hepatitis B core antibody or hepatitis B surface antigen must have a negative polymerase chain reaction (PCR) result before enrollment. Those who are PCR positive will be excluded.
* 11. Any uncontrolled active systemic infection.
* 12. Major surgery ≤ 4 weeks of first dose of study drug.
* 13. Any life-threatening illness, medical condition, or organ system dysfunction that, in the investigator's opinion, could compromise the subject's safety or put the study outcomes at undue risk.
* 14. Currently active, clinically significant cardiovascular disease, such as uncontrolled arrhythmia or Class 3 or 4 congestive heart failure as defined by the New York Heart Association Functional Classification; or a history of myocardial infarction, unstable angina, or acute coronary syndrome within 6 months prior to randomization.
* 15. Unable to swallow capsules or malabsorption syndrome, disease significantly affecting gastrointestinal function, or resection of the stomach or small bowel, symptomatic inflammatory bowel disease or ulcerative colitis, or partial or complete bowel obstruction.
* 16. Concomitant use of warfarin or other Vitamin K antagonists.
* 17. Receipt of a strong cytochrome P450 (CYP) 3A inhibitor within 7 days prior to the first dose of ibrutinib or requirement for continuous treatment with a strong CYP3A inhibitor.
* 18. Chronic liver disease with hepatic impairment Child-Pugh class B or C.
* 19. Lactating or pregnant.
* 20. Unwilling or unable to participate in all required study evaluations and procedures.
* 21. Unable to understand the purpose and risks of the study and to provide a signed and dated informed consent form (ICF) and authorization to use protected health information (in accordance with national and local subject privacy regulations).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Based on biological gender
Enrollment: 34 (Actual)
Dates: Start 2017-11-29 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Phase I: Maximum Tolerated Dose | 24 months
  Highest dose of ibrutinib from Phase 1 (420, 560, or 840 mg by mouth daily) that had fewer than two dose-limiting toxicities in its respective cohort
Phase II: Clinical Benefit Rate | 24 months
  To define the clinical benefit rate (CBR = CR [complete response] + PR [partial response] + SD [stable disease] > 6 months) of ibrutinib plus trastuzumab in patients with HER2-amplified, T-DM1-pretreated MBC

SECONDARY OUTCOMES:
Objective Response Rate | 24 months
  To determine the objective response rate (ORR = CR + PR) associated with ibrutinib plus trastuzumab.
Median Overall Survival | 24 months
  To assess median overall survival (OS) associated with ibrutinib plus trastuzumab.
Median Progression-free Survival | 24 months
  To assess median progression-free survival (PFS) associated with ibrutinib plus trastuzumab
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] of ibrutinib plus trastuzumab. | 24 months
  Number of Adverse Events and Serious Adverse Events from informed consent signature to 30 days after last dose of study drug, using Common Terminology Criteria for Adverse Events version 4.0 (CTCAE v4.03: June 14, 2010)
Pharmacokinetic Analysis for Ibrutinib (Phase I only)- Cmax | 24 months
  maximum (or peak) serum concentration that Ibrutinib achieves in Cycle 1 at indicated time points, and on Day 1 of cycle 3 for pharmacokinetic analysis
Pharmacokinetic Analysis for Ibrutinib (Phase I only)- Area under Curve | 24 months
  Area Under the Curve of Ibrutinib in 24 hours

OTHER OUTCOMES:
Cytokine Gene Expression Analysis | 24 months
  Changes in Th1- and Th2-related cytokine gene expression in whole blood, from Baseline to Week 12 to End of Treatment with ibrutinib plus trastuzumab, using NanoString human immunology gene panel.

CONTACTS AND LOCATIONS:
Overall Officials: Joyce O'Shaughnessy, MD, Principal Investigator — US Oncology Research/McKesson Specialty Health
Locations (1):
- 10 sites incl TX, WA, VA, and NV, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided